CLINICAL TRIAL: NCT05101083
Title: Speech Intelligibility in Quiet and Noise for New Versus Legacy Hearing Aids
Brief Title: Speech Intelligibility in Quiet and Noise for New vs. Legacy Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Starkey Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PR 21001
Record Dates: First submitted 2021-10-18; First posted 2021-11-01 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Crossover Assignment - Each participant will experience both test conditions (counterbalanced)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Hearing Aid 1 (Experimental): New Receiver-in-Canal device, successor of previous device generation
  Interventions: Device: Legacy Receiver-in-Canal Device
- Hearing Aid 2 (Active Comparator): Legacy Receiver-in-Canal device that is currently available on the market
  Interventions: Device: New Receiver-in-Canal Device

INTERVENTIONS:
Device: New Receiver-in-Canal Device — Successor of previous device generation
  Arms: Hearing Aid 2
Device: Legacy Receiver-in-Canal Device — Receiver-in-canal device available on the market
  Arms: Hearing Aid 1

SUMMARY:
This clinical investigation is designed to compare audiological performance (i.e., measurements of sound quality and speech understanding) between Starkey's new receiver-in-canal device and a commercially available legacy receiver-in-canal device.

DETAILED DESCRIPTION:
Starkey is investigating a new hearing aid with several new audiological features. These features have been assessed for benefit, individually, but this clinical investigation will serve as a test for safety and efficacy with all hearing aid features, together. The design of this study is a single-blinded, crossover design and will be conducted at Starkey's headquarters in Eden Prairie, MN.

ELIGIBILITY:
Inclusion Criteria:

* Adults, minimum age of 18
* Native English speakers
* Ability to complete questionnaires and laboratory assessments
* Symmetric, mild to moderately-severe sensorineural hearing loss
* Informed consent completed with signature

Exclusion Criteria:

* Inability to visit the Starkey Headquarters building for testing
* Central or middle ear hearing problems
* Medical contraindications to wearing hearing aids
* Learning disability, major cognitive handicap, or serious neurological or psychiatric disease that would prevent or restrict participation, as determined by the PI or designee

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility (% words repeated back correctly) in quiet and noise for new vs. legacy hearing aids | Four weeks
  IEEE sentences will be presented to the research participants in quiet and in background noise. The percent words repeated back correctly will be scored and serve as the reported result of this outcome measure.

SECONDARY OUTCOMES:
First fit ratings of sound quality on subjective questionnaires for the new vs. legacy hearing aids | Four weeks
  This data will be collected through lab testing following the first fit of the hearing aids. Participants will answer questionnaire items related to their impressions of sound quality. Results will be collected using a 7-point Likert scale, and ratings (1-7) will be analyzed using descriptive statistics. Statistical measures for repeated measurements will be used to understand any differences between hearing aid conditions.
Safety of the new, receiver-in-canal devices through tracking of adverse events | Four weeks
  This data will be collected through the tracking of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Starkey, Eden Prairie, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No